CLINICAL TRIAL: NCT05530304
Title: Outcome of a Triple Inner Branched Aortic Arch Stentgraft. A Prospective, Multicenter Registry.
Acronym: triple_branch
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Alexander Oberhuber, Univ.-Prof. Dr. med., University Hospital Muenster
Other Study IDs: University_Hospital_Muenster
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Aortic Arch; Aortic Arch Aneurysm; Dissection of Aortic Arch; Triple Branch
Keywords: Aortic arch pathologies; Aortic arch aneruysm; Aortic arch dissection; triple branch; stentgraft; Double branch; Inner branch
MeSH Terms: conditions — Aneurysm, Aortic Arch; Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Triple inner branched arch stentgraft — New findings regarding treatment planning and management of patients with aortic arch pathologies.

SUMMARY:
Outcome of a triple inner branched aortic arch stentgraft. A prospective, mulitcenter registry.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Presence of Aortic arch pathology
* Treatment planned with triple inner branch from Terumo Aortic
* Availability of the patients during the follow up period
* Informing patients about the study and providing written informed consent

Exclusion Criteria:

* Women of childbearing age
* Patients under 18 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited from patients presenting to participating hospitals with aortic pathology and meeting inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days after intervention
feasibility in terms of cannulation and stentgrafting of the three branches | During intervention
Stroke | 30 days after intervention

SECONDARY OUTCOMES:
Morbidity | during the follow up period of 3 year
  Access issue, paraplegia, kidney failure
Endoleaks Type I and III | during intervention and the follow up period of 3 year
Longterm mortality | during the follow up period of 3 year
Patency rate of branches | during the follow up period of 3 year
  primary and secondary
Stroke | during the follow up period of 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Oberhuber, MD, PhD, Study Chair — Department of Vascular and Endovascular Surgery University Hospital Münster
Locations (1):
- Muenster University Hospital, Münster, Germany